CLINICAL TRIAL: NCT06266507
Title: Examining the Effect of Occupational Therapy-Based Parent Coaching on Feeding Problems in Children With a History of Premature Birth
Brief Title: Examining the Effect of Occupational Therapy-Based Parent Coaching on Feeding Problems in Children With a Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Rukiye Begüm KOCA, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 169
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Feeding Behavior; Mother-Child Relations; Feeding and Eating Disorders
Keywords: prematurity; feeding problems; occupational therapy; parent coaching
MeSH Terms: conditions — Feeding Behavior; Feeding and Eating Disorders; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): Mothers who will receive a 10-week occupational therapy-based parent coaching intervention will be included in this group.
  Interventions: Behavioral: Ergotherapy Based Parent Coaching
- Control Group (Other): The control group will not receive an active intervention, but will be provided with an informative brochure on early childhood development. Additionally, once the research is completed, the right to participate in the intervention will be granted.
  Interventions: Other: Informative Brochure Distribution

INTERVENTIONS:
Behavioral: Ergotherapy Based Parent Coaching — Occupational Therapy Based Parent Coaching intervention will last 10 sessions and will be carried out on the online platform. Sessions are planned to last between 45-60 minutes. The interviews to be held during the sessions are considered as the basic principles of parent coaching; It will be carried out in line with the principles of joint planning, observation, implementation, reflection and feedback. This intervention aims to educate mothers on proper feeding strategies for their children and to enable them to carry out these practices independently.
  Other Names: Informative Brochure Distribution
  Arms: Research Group
Other: Informative Brochure Distribution — No active intervention will be made to the mothers in the target group; an informative brochure about early childhood development will be distributed.
  Arms: Control Group

SUMMARY:
Feeding problems are common in children with a history of premature birth, and these problems continue into early childhood. Feeding problems are affected by many biopsychosocial factors, and the context in which feeding takes place and the attitudes and behaviors of parents can also be effective in the emergence or continuation of these problems. The aim of our study is to evaluate the effects of occupational therapy-based parent coaching intervention on mothers and their children, who are considered to be primarily responsible for the feeding of children in our country. 46 mothers with premature children will be included in our study and participants will be randomly assigned to intervention/control groups. Mothers will fill out a sociodemographic information form, Canadian Occupational Therapy Measure (COPM), Behavioral Pediatric Feeding Assessment Scale, Sensory Profile Questionnaire - Oral Sensory Processing Subtest, Family Feeding Strategies Scale and Parental Self-Efficacy Scale via Google forms. Mothers in the research group will be given online occupational therapy-based parent coaching training for 10 weeks. Second evaluations will be carried out after the training; Final evaluations will be applied after 1 month of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity of the child (Birth week <37)
* The child is between 3-6 years old
* The mother must have the competence to use online platforms, technological tools and internet connection.
* The mother must have sufficient education to read, understand and fill out the scales.
* Mothers reporting complaints about feeding problems in their children

Exclusion Criteria:

* It may affect the child's feeding; Having a food allergy, disability, neurodevelopmental disease, chromosomal or structural anomalies
* The child is fed non-orally
* Being receiving occupational therapy, oral motor therapy or nutritional therapy at any center
* Not allowing practices such as video sharing, camera/audio sharing, and recording of sessions during the intervention.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Our intervention is aimed at mothers of children with a history of premature birth.
Enrollment: 39 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Behavioral Pediatric Feeding Assessment Scale | The scale will be applied 3 times in total: at the beginning of the study, 10 weeks after the first evaluation and 4 weeks after the second evaluation.
  This scale will be used to evaluate children's nutritional problems. Behavioral Pediatrics Feeding Assessment Scale (BPFAS) was developed by Crist and Napier Philips in 2001 and its original version consists of 35 questions. The usage age range of the survey is between 9 months and 7 years, and it is the scale with the most comprehensive reliability and validity data among the nutrition surveys administered by parents for preschool children. The questionnaire has good test-retest reliability and internal consistency, acceptable-to-good sensitivity, and good-to-excellent specificity. The BPFAS is capable of screening for a broad spectrum of feeding difficulties (nutritional and textural selectivity, food refusal, and oral motor difficulties). Turkish validity study by Önal et al. It was made by in 2017.
Sensory Profile Questionnaire - Oral Sensory Processing Test | The scale will be applied 3 times in total: at the beginning of the study, 10 weeks after the first evaluation and 4 weeks after the second evaluation.
  This scale will be used to examine how children's oral sensory processing skills change before and after the intervention. Ergotherapist Prof. Sensory Profile of the individual developed by Winnie Dunn; It is a measurement tool used to evaluate sensory modulation, in other words, the tendency to respond to sensory stimuli during daily activities and which sensory systems affect daily life more. It is used in children between the ages of 3-10. The individual; The test, which is used to measure functional performance in daily living activities, sensory processing abilities and sensory processing effects, consists of 3 main sub-parameters (sensory processing, modulation and behavioral-emotional responses) and 9 factor scores consisting of these parameters.
  *In our study, it was decided to use only the oral sensory processing subtest of questionnaire.
Canadian Occupational Therapy Measurement (COPM) | The scale will be applied 3 times in total: at the beginning of the study, 10 weeks after the first evaluation and 4 weeks after the second evaluation.
  The Canadian Occupational Performance Measurement (COPM) is an outcome measure designed to identify changes in individuals' perceived performance and satisfaction levels over time in the areas of self-care, productivity, and leisure. In the application of the COPM, the client is first interviewed and listed occupations they want to do, are expected to do, but are unable to do, or are dissatisfied with the way they are performed. Performance and satisfaction levels are recorded before and after the intervention, allowing the difference between the two assessments to be calculated. The COPM will be used in this study to determine participants' goals for the intervention and to examine changes in performance and satisfaction following the intervention for the identified occupations.

SECONDARY OUTCOMES:
Feeding Strategies Quesstionnaire | The scale will be applied 3 times in total: at the beginning of the study, 10 weeks after the first evaluation and 4 weeks after the second evaluation.
  This questionnaire will be used to measure whether mothers' feeding strategies have changed before and after the intervention.It is a scale developed by Berlin et al. in 2005 to measure parents' feeding strategies for their children. FSQ consists of 27 items and is administered to children between the ages of 2-6. FSQ; It consists of 6 subheadings: child control in eating, meal time, environment structure, family control in eating, release and coercive interventions. The FSQ scale includes answers ranging from 1 (strongly disagree) to 5 (strongly agree).
  It has been reported that the Feeding Strategies Scale can be used to evaluate child and parent feeding strategies regarding the prevention or treatment of pediatric feeding difficulties.
  A Turkish adaptation study was carried out by Meral in 2017, and the total Cronbach alpha value of the scale is 0.80.
Parental Self-Efficacy Scale | The scale will be applied 3 times in total: at the beginning of the study, 10 weeks after the first evaluation and 4 weeks after the second evaluation.
  This scale will be used to examine how parents' self-efficacy changes before and after parent coaching intervention. Parental Self-Efficacy Scale Guimond et al. It was developed by Cavkaytar et al. in 2005 and adapted into Turkish by Diken in 2007. It is a scale updated in 2014 and used to measure the self-efficacy perceptions of parents of children with disabilities regarding their parenting skills.
  The scale is a 7-point Likert-type rating scale and consists of a total of 17 items. The lowest score can be obtained from the scale, 17 points, and the highest score can be 119 points. As the score obtained from the scale increases, the level of self-efficacy also increases.
  Cronbach's Alpha internal consistency coefficient of the scale was found to be 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçen Akyürek, Ph. D., Study Director — Hacettepe University
Locations (1):
- Ankara Medipol University, Ankara, Ankara/ Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walton K, Daniel AI, Mahood Q, Vaz S, Law N, Unger SL, O'Connor DL. Eating Behaviors, Caregiver Feeding Interactions, and Dietary Patterns of Children Born Preterm: A Systematic Review and Meta-Analysis. Adv Nutr. 2022 Jun 1;13(3):875-912. doi: 10.1093/advances/nmac017. PMID 35157009
- [Background] Dev DA, Padasas I, Hillburn C, Stage VC, Dzewaltowski DA. Ecological Approach to Family-Style, Multilevel Child Care Intervention: Formative Evaluation Using RE-AIM Framework. J Nutr Educ Behav. 2022 Aug;54(8):728-744. doi: 10.1016/j.jneb.2022.03.005. Epub 2022 Jun 26. PMID 35768329